CLINICAL TRIAL: NCT04615338
Title: Outcomes and Trauma Pattern in Penetrating Neck Injuries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ezzat Mohamed Saleh, Physician, Assiut University
Other Study IDs: Open neck injuries
Record Dates: First submitted 2020-10-27; First posted 2020-11-04 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Neck Injuries
MeSH Terms: conditions — Neck Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Homicidal group: The group of patients presented with homicidal open neck injuries
  Interventions: Other: no intervension
- Suicidal group: The group of patients presented with suicidal open neck injuries
  Interventions: Other: no intervension
- Accidental group: The group of patients presented with accidental open neck injuries
  Interventions: Other: no intervension

INTERVENTIONS:
Other: no intervension — no intervention needed just observation and description

SUMMARY:
It is an observational retrospective multicenter study

DETAILED DESCRIPTION:
It is an observational descriptive, retrospective study. The study will be conducted in two centers: the Emergency and accident unit and Head and neck surgical unit Manchester Royal infirmary, Manchester, United Kingdom and Trauma unit and Otolaryngology department Assiut university Hospital, Assiut, Egypt. The study will include all the patients presented to both centers with open neck trauma in duration between April 2018 and October 2020. The following items recorded: gender, age, type of trauma (whether it is homicidal, suicidal, accidental trauma), time of the day the patients presented, Previous philological disorder in patients with suicidal types of trauma, number of neck wounds, site of the wounds ( in relation to the zones of the neck), size of each wound in centimeter, whether the wounds are deep or superficial to platysma, length of stay in the hospital, , injuries to any neck structures injuries in other parts of the body, involvement of other teams in management of the patent and type of involvement. Also the need of airway support (either intubation or tracheostomy), immediate and long term complications of the injury and if the patients needed neck exploration or just suturing of the wounds under local anesthesia.

Data of the patients who needed exploration will be reviewed to detect finding in neck exploration and try to find out the criteria of the patients who needed neck exploration and put a clear protocol for management.

The included patients will be categorized into 3 groups according to type of trauma (suicidal, homicidal or accidental) all the recorded data will be compared to detect the outcomes in each type of trauma and if there is a specific pattern of trauma in each category.

The study will be conducted after obtaining an institutional review board (IRB) approval from the committee of medical ethics, faculty of medicine, Assiut University. The study and all interventions and surgical procedures within it were done by scientifically qualified and trained personnel. The is no additional risk for participating in the study as it is a descriptive study

ELIGIBILITY:
Inclusion criteria:

1) All age groups regardless of sex. 2) Homicidal, suicidal and accidental type of trauma. 3) Patients with penetrating neck injuries due to sharp objects trauma. 4) Poly trauma patients having multiple body trauma as well as neck trauma will be included.

b. Exclusion criteria:

1. Patients with blunt neck trauma even if causing open wounds
2. Patients with neck burns
3. Patients with previous neck surgeries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients presented with open neck injuries regardless the cause of injury then will be categorized in to 3 groups according to the cause of trauma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
compare duration of the stay in the hospital in different types of open neck injuries | 1 year
  Duration of the stay of the patient in the hospital in days
compare fate of trauma in different types of open neck injuries | 1 year
  The fate of the trauma if the patient survived or died and if survived with long term complication
compare Site of wounds in different types of trauma | 1 year
  Site of wounds ( in which zone of the neck 1,2,3)
compare Number of wounds | 1 year
  Number of wounds
compare length of wound in different types of trauma | 1 year
  Length of each wound in cm
compare depth of wounds in different types of trauma | 1 year
  depth of each wound ( superficial or deep to platysma)
compare number of wound outside the neck i | 1 year
  Number of wounds outside the neck
Collect finding in neck exploration | 1 year
  Colect the finding that were found in neck exploration surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed EM Saleh, MSc, Principal Investigator — Assiut University
Locations (2):
- Assiut University Hospital, Asyut, Egypt
- Manchester royal infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided